CLINICAL TRIAL: NCT04313335
Title: Prophylactic Duloxetine Administration During Acute Herpes Zoster Prevents Postherpetic Neuralgia
Brief Title: Duloxetine for PHN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: China-Japan Friendship Hospital (Other); Tianjin Medical University Second Hospital (Other); Taiyuan Central Hospital of Shanxi Medical University (Other); Linfen Fourth People's Hospital (Unknown); Shandong Provincial Hospital (Other Government); Qingdao Municipal Hospital (Group) (Unknown); The Second People's Hospital of Huai'an (Other); First Hospital of China Medical University (Other); Second Affiliated Hospital of Zhengzhou University (Other); Fujian Provincial Hospital (Other); Cangzhou Central Hospital (Other); The People's Hospital of Fujian Province (Unknown); Beijing Tsinghua Chang Gung Hospital (Other); Peking University International Hospital (Other); Tianjin First Central Hospital (Other); Tianjin Huanhu Hospital (Other); Baoding First Central Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY 2020-009-02
Record Dates: First submitted 2020-03-07; First posted 2020-03-18 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Postherpetic Neuralgia
Keywords: Postherpetic Neuralgia, Duloxetine
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome of the study will be assessed by a third-party organization who will be blinded to the study allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine (Experimental): Apart from the standard treatment, participants in the Duloxetine Arm will be administered with oral duloxetine (up to 60 mg per day) in the acute herpes zoster period.
  Interventions: Drug: Duloxetine
- Control (No Intervention): Participants will be given the standard treatment during the acute herpes zoster period.

INTERVENTIONS:
Drug: Duloxetine — Oral Duloxetine (up to 60 mg per day) will be given, titrated, tapered in accordance with the pain intensity during the acute herpes zoster period.
  Arms: Duloxetine

SUMMARY:
In this study, the investigators aim to investigate the preventive efficacy of prophylactic oral duloxetine during acute herpes zoster on postherpetic neuralgia and its safety.

DETAILED DESCRIPTION:
Postherpetic neuralgia is a common complication of herpes zoster. Several interventions have been investigated for the treatment of postherpetic neuralgia, however, there is a lack of preventive intervention on postherpetic neuralgia. A recent retrospective study revealed that the administration of gabapentin during the acute herpes zoster period significantly decreased the incidence of postherpetic neuralgia. In the present study, the investigators aim to conduct a prospective, randomized, open-label, endpoint blinded study to investigate the preventive efficacy of prophylactic use of duloxetine on postherpetic neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* ages more than 50 years;
* diagnosed with uncomplicated acute herpes zoster;
* presents with vesicles within 72 hours;
* has an average pain score of at least 40/100 mm on a visual analog scale (VAS, 0 = no pain, 100 = worst possible pain, at opposite ends of a 100-mm line).

Exclusion Criteria:

* refuses to participate or to provide written informed consent;
* Zung Self-Rating Depression Scale raw score of more than 50 points;
* herpes zoster that involves with head, neck, ocular, mucous membrane, cranial nerve, or central nervous system;
* has hemorrhagic or necrotizing lesions, satellite lesions, abnormal vesicles or acute retinal necrosis;
* has been on immunosuppressive therapy or mono- or multi-pharmacotherapy that involves any tricyclic antidepressant, valacyclovir, duloxetine or cytotoxic medications before acute HZ onset;
* has been diagnosed with hepatic, renal or immune dysfunction;
* during pregnancy or breastfeeding at the time;
* hypersensitivity to the study drugs;
* has contraindications to valacyclovir or duloxetine;
* HZ vaccinated.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Preventive efficacy of Postherpetic neuralgia | 12 weeks after the reactivation of acute herpes zoster
  The proportion of participants in the Interventional Arm who gain a 0 score in a 100 mm visual analgue scale (0 mm = no pain, 100 mm = the most imaginable pain)

SECONDARY OUTCOMES:
Averaged weekly VAS score | up to 12 weeks
  Averaged weekly VAS score of each participant
Averaged weekly analgesic consumption | up to 12 weeks
  Averaged weekly consumption per analgesic of each participant
Patients' overall quality of life | At the end of Weeks 4, 8, and 12
  12-item Short-Form Health Survey (SF-12)
Sleep quality | At the end of Weeks 4, 8, and 12
  Pittsburgh Sleep Quality Index (PSQI) self-rated questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Drolet M, Brisson M, Schmader K, Levin M, Johnson R, Oxman M, Patrick D, Camden S, Mansi JA. Predictors of postherpetic neuralgia among patients with herpes zoster: a prospective study. J Pain. 2010 Nov;11(11):1211-21. doi: 10.1016/j.jpain.2010.02.020. PMID 20434957
- [Background] Johnson RW, Rice AS. Clinical practice. Postherpetic neuralgia. N Engl J Med. 2014 Oct 16;371(16):1526-33. doi: 10.1056/NEJMcp1403062. No abstract available. PMID 25317872
- [Background] Schutzer-Weissmann J, Farquhar-Smith P. Post-herpetic neuralgia - a review of current management and future directions. Expert Opin Pharmacother. 2017 Nov;18(16):1739-1750. doi: 10.1080/14656566.2017.1392508. Epub 2017 Oct 26. PMID 29025327
- [Background] Bulilete O, Leiva A, Rullan M, Roca A, Llobera J; PHN Group. Efficacy of gabapentin for the prevention of postherpetic neuralgia in patients with acute herpes zoster: A double blind, randomized controlled trial. PLoS One. 2019 Jun 5;14(6):e0217335. doi: 10.1371/journal.pone.0217335. eCollection 2019. PMID 31166976
- [Background] Ghanavatian S, Wie CS, Low RS, Zhang N, Montoya JM, Dhaliwal GS, Swanson DL. Premedication With Gabapentin Significantly Reduces the Risk of Postherpetic Neuralgia in Patients With Neuropathy. Mayo Clin Proc. 2019 Mar;94(3):484-489. doi: 10.1016/j.mayocp.2018.11.004. Epub 2019 Feb 2. PMID 30718068
- [Derived] Zhao C, Zhang T, Zhu Q, Chen Z, Ren H, Shrestha N, Meng L, Shen Y, Luo F. PROCESS Trial: Effect of Duloxetine Premedication for Postherpetic Neuralgia Within 72 Hours of Herpes Zoster Reactivation-A Randomized Controlled Trial. Clin Infect Dis. 2024 Apr 10;78(4):880-888. doi: 10.1093/cid/ciad714. PMID 38015658
- [Derived] Chen Z, Shrestha N, Zhao C, Fan B, Luo F. Effect of duloxetine premedication for postherpetic neuralgia within 72 h of herpes zoster reactivation [PROCESS]: a study protocol for a randomized controlled trial. Trials. 2020 Dec 9;21(1):1012. doi: 10.1186/s13063-020-04919-6. PMID 33298154